CLINICAL TRIAL: NCT06602284
Title: A Full Face, Baseline Controlled Study to Evaluate the Efficacy of Dermapen 4™ Microneedling Device in Conjunction with MG-CLR Serum for Acne Treatment Over 12 Weeks.
Brief Title: A Full Face Study to Evaluate the Efficacy of Dermapen 4™ Microneedling Device in Addition with MG-CLR Serum for Acne Treatment Over 12 Weeks.
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Equipmed USA LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SKIN/EMAC/2024-01
Record Dates: First submitted 2024-09-16; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acne
Keywords: dermapen, microneedling, acne
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- A single arm, full face clinical study. (Other): Dermapen 4 in conjunction with MG-CLR serum
  Interventions: Combination Product: Dermapen 4™

INTERVENTIONS:
Combination Product: Dermapen 4™ — Dermapen 4™ conjunction with MG-CLR

SUMMARY:
This study is conducted to check how well the Dermapen 4™ microneedling device works with MG-CLR serum for treating acne over 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects aged between 18-45 years (both ages inclusive)
2. Fitzpatrick skin phototype I to VI.
3. Subjects having IGA score of 2 and 3.
4. Subjects who have not received any kind of treatment for acne 1 month before the start of the study.
5. Subject free of excessive hair, cuts, abrasions, fissures, wounds, lacerations, or any other skin conditions on the face.
6. Subjects who agree not to use any other product/treatment/home remedy/ except the provided products on their face during the study period

Exclusion Criteria:

1. Subjects with known skin condition that may impact the assessment.
2. Subjects with active Herpes labialis infection.
3. Subjects known to have bleeding and clotting disorders (self-declared).
4. Subjects known to have connective tissue disorders.
5. Subjects with any other signs of significant local irritation or skin disease.
6. Subjects currently taking any medication, which the investigator believes may influence the interpretation of the data.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 10 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Acne severity | 13 weeks
  Change in acne severity using the modified GAGS scale at all time points when compared to baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Skin Wellness Dermatology, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: protocol will be available soon after approval
Access Criteria: Sponsor and CRO/site personals